CLINICAL TRIAL: NCT06737302
Title: Epidemiology (and Natural History) of Sleep Disordered Breathing and Respiratory Support in Children and Young People With Cerebral Palsy
Brief Title: Epidemiology of Sleep Disordered Breathing in Children and Young People With Cerebral Palsy
Acronym: UK_CPSSS
Status: Recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: AC24189
Record Dates: First submitted 2024-12-06; First posted 2024-12-17 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Palsy (CP); Sleep Disordered Breathing (SDB); Respiratory Support
Keywords: sleep disordered breathing; cerebral palsy; respiratory support
MeSH Terms: conditions — Cerebral Palsy; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cerebral palsy (CP) refers to a non-progressive movement disorder, which occurs due to damage to the developing brain around the time of birth. Symptoms of sleep disordered breathing (SDB) include noisy breathing during sleep,increased day-time sleepiness and reduced energy levels. In the long term, SDB might have an effect on the brain and learning, as well as putting strain on the heart.

Children with CP have a higher risk of sleep breathing problems compared to typically-developing children, and the negative impact of sleep disturbance in children with CP on their family members/carers' sleep and mental health cannot be understated. Early recognition and management of SDB is important for children with CP to give these children the best possible sleep quality, and to maximise learning potential.

SDB in children with CP is often under-recognised and under-treated. Treatment of SDB in children with CP might involve wearing a mask that delivers pressurised air to hold open a child's airway and make breathing easier when they are asleep. This is called 'respiratory support' which can be continuous pressure (CPAP) or non-invasive ventilation (NIV) which is pressure support with a back-up breathing rate. There is limited knowledge on the appropriate indications or timing to use them.

Though respiratory support in children with CP is proven to help with breathing during sleep, its impact on quality of life, number of hospital admissions or frequency of chest infections is unknown.

This study will look at the number of children with CP on respiratory support across the UK, as well as the number of children newly diagnosed with SDB and/or established on respiratory support over a 1-year period. This study will also explore socioeconomic factors that might influence access of sleep services and the perceived facilitators and barriers to successfully initiating respiratory support in children with CP.

DETAILED DESCRIPTION:
The study will be conducted as a nationwide UK Sleep Surveillance Survey of children with cerebral palsy. It will be conducted as a two-part survey (UK-wide point prevalence survey and UK-wide Incidence self-reporting form).

There is no national registry of children with cerebral palsy (CP) which collects information on sleep or sleep disordered breathing (SDB) for the purpose of this study. Hence, the investigators will recruit all tertiary paediatric centres across the UK which offers sleep services to children. A single point of contact will be identified for further communication and to act as local champion for collecting the relevant information in each centre.

I) National point prevalence survey;

* Single point of contact (PoCo) identified across tertiary paediatric centre which offer sleep services
* Single questionnaire sent on pre-specified date to PoCo in each centre
* Study will aim to;

  * assess number of children in each centre with CP established on respiratory support
  * gather information on practices in different centres pertaining to their assessment and management of children with CP and suspected SDB

II) National Incidence self reporting form;

* This phase of the review will a conducted over a 1-year period
* Will be conducted as a 2-part survey, with the PoCo being sent a monthly self-reporting form;

  * Part A;

    * To identify number of children with CP who underwent sleep study, the proportion of those who were diagnosed with SDB, and the total number of children with CP who were initiated on respiratory support (regardless of sleep study results) in that calendar month
    * To be completed by PoCo in all centres
    * If any children with CP were newly initiated on respiratory support (regardless of sleep study results), PoCo will be directed to complete Part B
  * Part B;

    * Will gather further information on children with CP who were initiated on respiratory support in the calendar month (regardless of sleep study results), with a separate form for each child
    * Data collected will assess association between socio-economic factors (ethnicity, social deprivation index and urban-rural classification) and diagnosis of sleep disordered breathing and/or being initiated on respiratory support in children with CP
* No power calculation has been done for this review, as this is an observational study with an aim to include all children with cerebral palsy, newly diagnosed with SDB and/or started on respiratory support in the UK

ELIGIBILITY:
Inclusion Criteria:

Cases for Prevalence survey;

* Any child aged ≤16 years old, with a confirmed diagnosis of cerebral palsy
* On respiratory support on the date of prevalence survey

Cases for Incidence self-reporting form;

* Part A;

  * Any Child aged ≤16 years old, with confirmed diagnosis of cerebral palsy
  * Had sleep studies for suspected sleep disordered breathing within the preceding calendar month
* Part B;

  * Any Child aged ≤16 years old, with a confirmed diagnosis of cerebral palsy
  * Initiated respiratory support (CPAP or NIV or invasive tracheostomy ventilation) in the preceding month

Exclusion Criteria: (For prevalence survey and incidence self-reporting form)

* Any patient aged >16 years old
* Patient does not have a confirmed diagnosis of cerebral palsy

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: UK (England, Scotland, Wales and Northern Ireland)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Prevelance | Day 1 of study
  Identify the prevalence of children with cerebral palsy on respiratory support across the UK
Incidence | 13 months
  Identify the incidence of children with CP newly diagnosed with sleep disordered breathing across the UK

SECONDARY OUTCOMES:
Screening questionnaire | 13 months
  Type of questionnaire used for screening for SDB in children with CP
Types of sleep studies | 13 months
  Types of sleep studies used across the UK in investigating SDB in children with CP
Types of respiratory support | 13 months
  Types of respiratory support offered for managing SDB for children with CP
Indications for starting respiratory support | 13 months
  Quantify the indications for starting respiratory support in each child with CP
Social deprivation | 13 months
  Explore association between social deprivation and likelihood of accessing and/or initiating respiratory support for SDB
Ethnicity | 13 months
  Explore association between ethnicity and likelihood of accessing and/or initiating respiratory support for SDB
Geographical location | 13 months
  Visualization of regions with underrepresentation/reporting of children with CP needing respiratory support for SDB
Facilitators | 13 months
  Quantify perceived facilitators to successfully setting up and establishing respiratory support for SDB in children with CP
Barriers | 13 months
  Quantify perceived barriers to successfully setting up and establishing respiratory support for SDB in children with CP

CONTACTS AND LOCATIONS:
Locations (1):
- NHS Lothian, Edinburgh, Edinbrugh, United Kingdom

IPD SHARING:
Plan to Share IPD: No